CLINICAL TRIAL: NCT04665622
Title: Theory of Mind, Empathy and Eye Gaze Strategies During an Artwork Observation in Neurodegenerative Pathologies.
Brief Title: Assessment of Empathetic Process by Scanpath Study of an Artwork
Acronym: EYE-EMPATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: Association de Recherche Bibliographique pour les Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EYE-EMPATH
Record Dates: First submitted 2017-03-08; First posted 2020-12-11 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Dementia; Parkinson Disease; Fronto-Temporal Dementia
Keywords: Eye-Tracking; Empathy; Social cognition; Theory of Mind; Scanpath; Gaze
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A monocentric prospective, descriptive, comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fronto-temporal Dementia (Other): 10 subjects
  Interventions: Other: Eye-Tracking / Neuropsychological evaluations
- Alzheimer's Dementia (Other): 20 subjects
  Interventions: Other: Eye-Tracking / Neuropsychological evaluations
- Parkinson's Disease (Other): 20 subjects
  Interventions: Other: Eye-Tracking / Neuropsychological evaluations
- Healthy volunteers (Other): 20 subjects
  Interventions: Other: Eye-Tracking / Neuropsychological evaluations

INTERVENTIONS:
Other: Eye-Tracking / Neuropsychological evaluations — Use of Eye-Tracking / Neuropsychological évaluations in 4 groups

SUMMARY:
Analysis of gaze patterns during social cognition tasks and standardised exploration of a specific artwork, between elderly subjects without cognitive disorders and subjects with neurodegenerative diseases such as Fronto-Temporal Dementia, Alzheimer's Dementia or Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Male or Female.
* 60 years old and above.
* Sufficient written and oral expression in French.
* Benefit from French or Monaco Social security.
* Written informed consent signed by the patient.
* For the control group: voluntary subjects, without cognitive impairment.
* For the FTD / AD / PD groups: patients diagnosed with one of these diseases, and volunteers to participate in the study.

Exclusion Criteria:

* General anaesthesia within 3 months.
* Ophthalmological problems preventing a video-oculography examination.
* Oculomotor disorders such as "fixation disorders" or "ocular tracking disorders".
* History of stroke.
* Cognitive disorders of the type: visual agnosia, visuo-spatial disorder, visuo-perceptual disorder or aphasia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
1. Gaze patterns | baseline
  Comparison of gaze patterns between the control group and the pathological groups, during standardized exploration of a specific artwork. Evaluation criteria: difference in the number of fixation
2.Gaze Patterns | Baseline
  Comparison of gaze patterns between the control group and the pathological groups, during standardized exploration of a specific artwork. Evaluation criteria: difference in exploration strategy (chronology) on target areas.
3.Gaze Patterns | Baseline
  Comparison of gaze patterns between the control group and the pathological groups, during standardized exploration of a specific artwork. Evaluation criteria: difference in time spent on target areas.

SECONDARY OUTCOMES:
Cognitive Theory of mind during an artwork observation: Score 1 | Baseline
  Subject's estimation of the distance perceived by the character represented on the artwork, at a 1st and a 2nd observation of the painting. Score 1 is the ratio of estimated distances (distance2/distance1).
Cognitive Theory of mind during an artwork observation: Score 2 | Baseline
  Subject's estimation of the time perceived by the character represented on the artwork, at a 1st and a 2nd observation of the painting. Score 2 is the ratio of estimated times (time2 / time1).
Cognitive Theory of mind: TOM-15 a false-belief task to assess cognitive theory of mind | Baseline
  The task presents 15 stories. The subject must answer the question asked by choosing among two propositions, the correct answer consisting in attributing the correct belief to the character represented. Total score (/ 15).
  ToM 15 is used as reference test for correlation study with score1 and score 2.
Affective ToM (Score 3) | Baseline
  At observation, 1 and 2, subject must attribute an emotion to the character represented on the artwork, choosing an answer among 6 propositions: 3 negative mental states, 2 neutral and 1 positive.
  Score 3 rating : 2 points if a negative emotion is attributed to the 1st and 2nd observation; 1 point if the negative emotion is attributed only to the 2nd observation; 0.5 point if the negative emotion is attributed only to the 1st observation; 0 point if no negative emotion is attributed.
Affective ToM : The Reading the Mind in the Eye test - RME - (Baron-Cohen S at al., 2001) | Baseline
  The task consisted of 36 black-and-white photographs of the eye area of faces. Subject is asked to choose which word, among four options, best described what the character in the photograph was thinking or feeling. Total score (/36) and three emotional valence sub-scores: positive (/8), neutral (/16) and negative (/12) according to the procedure described by Harkness et al., 2005.
  RME is used as reference test for correlation study with Score 3.
Affective empathy: Score 4. | Baseline
  Intensity of the emotion felt by the participant following observation of the table, using an EVA scale [0-10].
Affective empathy: The Empathy Quotient (EQ). | Baseline
  Self-administered questionnaire of 40 questions. Participant must choose one of the four propositions ("strongly agree", "tend to agree", "tend to disagree", "strongly disagree") awarding 0, 1 or 2 points. Total Score / 60.
  EQ is used as reference test for correlation study with Score 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No